CLINICAL TRIAL: NCT04109300
Title: Pharmacogenomic Strategies in Inflammatory Bowel Disease: Evaluating the Role of Pre-emptive HLADQA1 Genotyping for the Application of Targeted Infliximab-based Combination Therapy (INHERIT)
Brief Title: Preemptive HLA Genotyping for the Safe Use of Infliximab-combination Therapy in Inflammatory Bowel Disease
Acronym: INHERIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HLAADA1
Record Dates: First submitted 2019-09-27; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
Keywords: Pharmacogenomics; Combination therapy; Infliximab
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to prospective HLADQA1*05A>G screening and targeted administration of combination therapy or standard of care (administration of combination therapy is at the discretion of the treating physician) and followed up to one year or until infliximab discontinuation. HLADQA1*05A>G genotyping will be performed in the standard of care group; however, investigators will remain blinded to this outcome until study completion.
Who Masked: Participant, Outcomes Assessor
Masking Description: This will be a single-blinded study. The treating gastroenterologist will be unblinded to the participant's allocation, while the assessor seeing the patient at the initial visit (PM Clinic) and at the subsequent follow up visits (week 14, week 26, week 52) will be blinded to the intervention (preemptive screening versus standard do care).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- preemptive screening (Experimental): prospective HLADQA1*05A>G screening and targeted administration of combination therapy of infliximab with one of either methotrexate or azathioprine.
  Interventions: Genetic: HLADQA1*05A>G screening
- standard of care (Active Comparator): administration of combination therapy with infliximab and one of methotrexate or azathioprine is at the discretion of the treating physician. HLADQA1*05A>G genotyping will be performed retrospectively.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Genetic: HLADQA1*05A>G screening — DNA will be extracted from whole blood collected from subjects in both arms using the MagNA Pure Compact instrument (Roche, Laval, Quebec, Canada). A custom TaqMan allelic discrimination assay (Applied Biosystems, Carlsbad, CA) will be used to determine the presence of wild-type and/or variant alleles in the class II HLA gene region at rs2097432 mapped to the HLA-DQA1*05 region in infliximab-exposed IBD subjects. Genetic data will be used to determine whether or not one of methotrexate or azathioprine should be applied to the patient in the experimental arm.
  Arms: preemptive screening
Other: Standard of Care — The treating physician will use clinical judgement to determine need for the addition of one of methotrexate or azathioprine to infliximab therapy.
  Arms: standard of care

SUMMARY:
Inflammatory bowel disease (IBD) is a common disease in Canada, leading to significant morbidity as a result of remitting and relapsing intestinal inflammation. Currently, tumor necrosis factor (TNF) antagonists such as infliximab, make up 30% of the biologic agents available to individuals with IBD. There is a high risk of losing response or having a hypersensitivity reaction to infliximab, necessitating treatment discontinuation. This is due, in part, to the formation of anti-drug antibodies (ADAs). ADA formation can result in loss of response to therapy which may eliminate an intestine-saving therapy and increases their risk of progressing to surgical resection. There are few tools clinicians can implement to minimize the risk of ADA formation. The current approach is to add a second drug (known as combination therapy), specifically an immunomodulator (methotrexate or azathioprine), exposing the patient to additional medication-related risks, intensive monitoring with bi-weekly blood work and potential side effects including infection and malignancy.

Preliminary data from our group as well as others suggests that individuals who carry a variant in the class 2 human leukocyte antigen (HLA) gene (HLADQA1*05A>G, rs2097432) are more likely to form ADAs to infliximab. Pre-emptive screening for this variant may allow clinicians to more selectively use combination therapy, recommending it only in IBD patients at high risk of developing ADAs to infliximab. Additionally, this may result in fewer drug-associated adverse events.

With this project, we aim to explore the value of prospective HLADQA1*05 screening (pharmacogenomic screening) in IBD patients being considered for treatment with infliximab and using the result to guide the application of combination therapy compared to IBD patients treated with infliximab (with or without a second agent) as per current practice. We will assess the incidence of infliximab ADA formation, as well as the incidence of infliximab loss of response, treatment discontinuation, and adverse drug events. Additionally, we will assess the time to each of these events.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) affects over 250,000 individuals in Canada. It is comprised of ulcerative colitis (UC) and Crohn's disease (CD). The dysregulated inflammatory response targeting the gastrointestinal (GI) tract is the hallmark of IBD and can lead to significant physical and psychological morbidity amongst affected individuals. Hallmarks of the disease include hematochezia, diarrhea, and abdominal pain. Individuals with IBD are committed to long-term immunosuppressive therapy to drive disease into remission; however, such treatments are associated with significant cost, as well as, a risk for significant drug-related toxicities. Individuals who are resistant or lose response to traditional therapies may require hospitalization and intestinal resection or colectomy. This is also associated with significant costs to the health care system and to patients.

The last decade has seen an expansion in the number of therapies, specifically monoclonal antibodies (biologics), available for the treatment of IBD, targeting and inhibiting different proteins involved in perpetuating the inappropriate inflammatory response. There is growing evidence to support the use of biologics early in the disease course, bypassing other less effective and older treatments. In Canada there are currently five biologic agents approved for the management of IBD: infliximab, adalimumab, golimumab, vedolizumab and ustekinumab. Infliximab, the first biologic approved for the management of IBD in Canada and the most widely used, is a chimeric human-murine monoclonal antibody directed against the pro-inflammatory cytokine, tumour necrosis factor-α (TNF). The efficacy of infliximab in CD and UC has been demonstrated in landmark trials; ACCENT and ACT respectively. It is considered a standard of care for moderate to severe IBD in treatment algorithms.

Unfortunately, up to 40% of patients who initially respond to a TNF antagonist such as infliximab will lose response by the one-year mark. Additionally, up to 23% of individuals with IBD exposed to infliximab will have an immediate infusion reaction with flushing, urticaria, presyncope and dyspnea necessitating treatment cessation. A leading contributor to both loss of response and infusion reactions is the development of anti-drug antibodies (ADAs).

ADAs are a consequence of the "immunogenicity" of TNF antagonists. Immunogenicity refers to the immune response of the exposed individual against large molecule therapeutic proteins such as infliximab. The underlying mechanisms of immunogenicity in TNF antagonist-exposed IBD patients are poorly defined. Clinically, ADAs are very relevant to IBD treatment as some ADAs can inhibit drug function or induce hypersensitivity in exposed patients. Studies have shown that the presence of ADAs correlates with a loss of response to infliximab as well as with a high risk of infusion reaction.

Therapeutic drug monitoring, the ability to measure ADAs, in addition to serum drug concentrations, has revolutionized IBD treatment algorithms by providing objective evidence to inform clinical decision-making. Unfortunately, the current tools are only able to identify ADAs once they have developed and thus, treatment adjustments are reactive as opposed to preemptive. Patients are often only screened for ADAs once loss of response or a hypersensitivity reaction have occured. One way clinicians attempt to reduce the risk of ADA formation is to empirically combine a second immune-suppressing agent such as methotrexate or azathioprine (immunomodulators) with infliximab. The addition of an immunomodulator to infliximab-based therapy (combination therapy) is associated with reduced ADA formation. The downside is that combination therapy may be associated with an increased risk of infection, malignancy and other side effects related to the immunomodulator (pancreatitis, myelotoxicity, hepatotoxicity). There is also concern over the use of dual immunosuppression in certain patient populations, including frail elderly or patients at high risk of infection or malignancy.

Currently, there are no clinical tools that predict who will develop ADAs, lose response to or have a hypersensitivity reaction to infliximab. Additionally, there are few ways to predict the risk of adverse events in IBD patients treated with combination therapy. Recently, in an peer-reviewed dataset, a group demonstrated that variation in the class 2 human leukocyte antigen (HLA) gene region (HLADQA1*05A>G, rs2097432) is linked to an increased risk of ADA formation against infliximab and to a lesser extent, its sister TNF-antagonist, adalimumab18. In a separate, retrospective study, we have confirmed that variation in HLADQA1*05A>G (rs2097432) is independently-associated with a significantly higher incidence of and faster progression to infliximab ADA formation. Moreover, we demonstrated that variant carriers had a higher risk of infliximab loss of response, treatment discontinuation as well as a faster progression to these outcomes (Wilson et.al. 2019 unpublished/Gastro, submitted). Interestingly, the addition of co-immunosuppression (methotrexate or azathioprine) to infliximab therapy reduced the risk of antibody formation in variant carriers compared to that of an individual with a wild type genotype.

Having the capacity to identify individuals at high risk of ADA formation and apply targeted combination therapy to those individuals and avoid combination therapy in others would be exceedingly valuable in clinical practice. Thus, we propose to assess the utility of preemptively screening patients with IBD who are being considered for infliximab therapy for HLADQA1*05A>G and applying co-immunosuppression with an immunomodulator (methotrexate or azathioprine) to the variant carriers (AG or GG) compared to those received the current standard of care. We will assess the resultant impact on infliximab ADA formation in addition to highly relevant clinical outcomes such as infliximab loss of response, treatment discontinuation, and adverse drug events.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>17 years of age) with a histopathologic diagnosis of CD or UC being initiated on therapy with infliximab by their treating gastroenterologist
* Individuals with prior biologic exposure to a non-TNF-based therapy are eligible
* Individuals on prednisone are eligible

Exclusion Criteria:

* Absence of histopathologic diagnosis of CD or UC
* Prior exposure to a TNF-based therapy (infliximab, golimumab, adalimumab)
* Pregnancy
* Known contraindication to both azathioprine and methotrexate
* Non-english speaking
* Being ineligible for infliximab based on insurance plan

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
incidence of infliximab anti-drug antibodies | 1 year
  Evaluate the impact of pharmacogenomic screening and the administration of targeted-combination infliximab therapy to high risk (variant-carrying) individuals compared to an unscreened IBD population receiving standard of care (where combination therapy is administered at the discretion of the physician) on the incidence of infliximab ADA formation. Infliximab ADA formation is defined as any detectable amount of ADA in the absence of detectable serum infliximab (measured by enzyme-linked immunosorbent assay, ELISA).

SECONDARY OUTCOMES:
incidence of infliximab loss of response | 1 year
  defined as a relapse in clinical symptoms after week 14 of infliximab dosing, with an increase in the Harvey Bradshaw index (HBI) ≥ 3 points or the partial Mayo score ≥ 3 points, following a response to infliximab induction therapy where a 3-point reduction was seen in the HBI or partial Mayo score
incidence of infliximab discontinuation | 1 year
  when stopped by treating physician
incidence of infliximab-related adverse drug events | 1 year
  defined as any injury presumed secondary to infliximab exposure as deemed by the treating gastroenterologist. This is including but not limited to: infection, immediate infusion reaction, delayed infusion reaction, psoriaform rash
incidence of immunomodulator-related adverse drug events | 1 year
  defined as any injury presumed secondary to azathioprine or methotrexate exposure as decided by the treating gastroenterologist. This is including, but not limited to: infection, nausea and dyspepsia, myelotoxicity, hepatoxicity, pancreatitis
incidence of combination therapy (infliximab and one of methotrexate or azathioprine) -related adverse drug events | 1 year
  defined in outcome 4 and 5
time to infliximab anti-drug antibody formation | 1 year
  measured from the time of treatment initiation to the time of antibody formation
time to infliximab loss of response | 1 year
  measured from the time of treatment initiation to the time of infliximab loss of response defined as a relapse in clinical symptoms after week 14 of infliximab dosing, with an increase in the Harvey Bradshaw index (HBI) ≥ 3 points or the partial Mayo score ≥ 3 points, following a response to infliximab induction therapy where a 3-point reduction was seen in the HBI or partial Mayo score.
time to infliximab discontinuation | 1 year
  measured from the time of treatment initiation to the time of cessation as decided by the treating physician.

CONTACTS AND LOCATIONS:
Overall Officials: Aze A Wilson, MD, PhD, Principal Investigator — Western University
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No